CLINICAL TRIAL: NCT05221034
Title: Cross-Cultural Adaptation, Reliability, Validity, and Responsiveness of the Urdu Version of Questionnaire for Female Urinary Incontinence Diagnosis
Brief Title: Urdu Version of Questionnaire for Female Urinary Incontinence Diagnosis: Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00283
Record Dates: First submitted 2022-02-01; First posted 2022-02-02 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Questionnaire for female Urinary Incontinence Diagnosis; Cultural adaptation; Validity; Urdu Version; Reliability; Pelvic Floor Distress Inventory
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study will be to translate and culturally adapt Questionnaire for Female Urinary Incontinence Diagnosis into the Urdu language and to evaluate its reliability and validity in the Pakistani urinary incontinence population. Also assess its correlation with Pelvic Floor Impact Questionnaire, Pelvic Floor Distress Inventory, International Consultation on Incontinence Questionnaire-short form for severity and also check the quality of life.

DETAILED DESCRIPTION:
According to the previous recommendation, Questionnaire for Female Urinary Incontinence Diagnosis will be translated into the Urdu language from its original English version and adapted culturally in Pakistan. Amongst the urinary incontinence population, Questionnaire for Female Urinary Incontinence Diagnosis will be distributed in 200 patients who would be recruited by a convenience sampling technique under the pre-defined inclusion and exclusion criteria after signing the informed consent forms. To test the inter-observer reliability and intra-observer reliability of the Pelvic Floor Impact Questionnaire, Pelvic Floor Distress Inventory, International Consultation on Incontinence Questionnaire-short form questionnaires will be completed by two observers, on the same day, with a time interval of 2 hours between first and second distribution. For the 3rd assessment, questionnaires will be completed after 7 days by the first observer, for intra-observer assessment. Statistical Package of Social Sciences software version 24 will be used for the purpose of data entry and analysis. Internal consistency will be analyzed by Cronbach alpha value. Test-retest reliability will be assessed by using an intra-class correlation coefficient. The Questionnaire for Female Urinary Incontinence Diagnosis will be evaluated for content validity, construct validity, criterion validity, and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 years or above.
* Women who answered 'yes' to one or both of the following questions: "In the last month have your urine leaked involuntarily when you lifted weights, exercised, sneezed or coughed?" and "In the last month, have you sensed very strong urge to urinate, leaking urine before getting into the bathroom?"

Exclusion Criteria:

* Current pregnancy or 3 months postpartum
* Any neurological disease
* Urinary tract infection, urogenital cancer, interstitial cystitis
* Taking treatment for PFD in the last 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — * Women age 18 years or above.
  * Women who answered 'yes' to one or both of the following questions: "In the last month have your urine leaked involuntarily when you lifted weight, exercised, sneezed or coughed?" and "In the last month, have you sensed very strong urge to urinate, leaking urine before getting to bathroom?"
Study Population: Pakistani women suffering from urinary incontinence.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Questionnaire for Urinary Incontinence Diagnosis | 1st day
  Questionnaire for Urinary Incontinence Diagnosis is a 6-item tool and its main purpose is to diagnose the two major kinds of urinary incontinence which are stress urinary incontinence and urge urinary incontinence. The first three questions of questions for Urinary Incontinence Diagnosis are related to stress and the next three are related to urge type. By totaling the response of each item the score of each domain is calculated and separated for both Stress Urinary Incontinence and Urgency Urinary Incontinence with the score of each ranging from 0 to 15. The cutoff value for Stress Urinary Incontinence is equal to or greater than 4 and the cutoff value for Urgency Urinary Incontinence is equal to or greater than 6
Pelvic Floor Distress Inventory | 1st day
  Pelvic Floor Distress Inventory consists of twenty questions which are divided into three subscales (Pelvic organ prolapse, intestine, and bladder portion)
Pelvic Floor Impact Questionnaire | 1st day
  Pelvic Floor Impact Questionnaire contains 7 questions with 3 domains (urinary, pelvic organ prolapse, and colon-rectal anal).
International Consultation on Incontinence Questionnaire-Short Form | 1st day
  International Consultation on Incontinence Questionnaire-Short Form is a valid tool to assess the severity and impact of urine incontinence on the quality of life in females. The International Consultation on Incontinence Questionnaire-Short Form is a six-item tool out of which four major items are asked for the symptoms of urinary incontinence that happen in the previous four weeks. Item 1 and 2 are the demographics whereas items 3,4,5 are asked for the actual score of urinary incontinence. item 6 is a self-analytical question for urinary incontinence type

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No